CLINICAL TRIAL: NCT03885011
Title: A Multi-Center, Double-Masked Evaluation of the Efficacy and Safety of CSF-1 in the Treatment of Presbyopia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Orasis Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-150-0006
Record Dates: First submitted 2019-03-19; First posted 2019-03-21 (Actual); Results first posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2022-09

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia | interventions — Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- CSF-1 (Experimental): This treatment arm consists of 2 different concentrations of CSF-1. Subjects randomized to the CSF-1 treatment arm will receive their first dose of CSF-1 in-office at Visit 2. All subjects will dose twice a day in both eyes with a single drop for approximately 1 week. At Visit 3, subjects randomized to the CSF-1 arm will now receive a different concentration of CSF-1. Subjects will continue dosing twice a day in both eyes for approximately 1 week.
  Interventions: Drug: CSF-1
- CSF-1 Component #1 (Active Comparator): This treatment arm consists of 2 different concentrations of CSF-1 Component #1.
  Subjects randomized to the CSF-1 Component #1 treatment arm will receive their first dose of CSF-1 Component #1 in-office at Visit 2. All subjects will dose twice a day in both eyes with a single drop for approximately 1 week. At Visit 3, subjects randomized to the CSF-1 Component #1 arm will now receive a different concentration of CSF-1 Component #1. Subjects will continue dosing twice a day in both eyes for approximately 1 week.
  Interventions: Drug: CSF-1 Component #1
- CSF-1 Component #2 (Active Comparator): This treatment arm consists of a single concentration of CSF-1 Component #2. Subjects randomized to the CSF-1 Component #2 treatment arm will receive their first dose of CSF-1 Component #2 in-office at Visit 2. All subjects will dose twice a day in both eyes with a single drop for approximately 1 week. At Visit 3, subjects randomized to the CSF-1 Component #2 arm will continue dosing with the same concentration of CSF-1 Component #2. Subjects will continue dosing twice a day in both eyes for approximately 1 week.
  Interventions: Drug: CSF-1 Component #2

INTERVENTIONS:
Drug: CSF-1 — This treatment arm consists of 2 different concentrations of CSF-1. Subjects randomized to the CSF-1 treatment arm will receive their first dose of CSF-1 in-office at Visit 2. All subjects will dose twice a day in both eyes with a single drop for approximately 1 week. At Visit 3, subjects randomized to the CSF-1 arm will now receive a different concentration of CSF-1. Subjects will continue dosing twice a day in both eyes for approximately 1 week.
  Arms: CSF-1
Drug: CSF-1 Component #1 — This treatment arm consists of 2 different concentrations of CSF-1 Component #1.
  Subjects randomized to the CSF-1 Component #1 treatment arm will receive their first dose of CSF-1 Component #1 in-office at Visit 2. All subjects will dose twice a day in both eyes with a single drop for approximately 1 week. At Visit 3, subjects randomized to the CSF-1 Component #1 arm will now receive a different concentration of CSF-1 Component #1. Subjects will continue dosing twice a day in both eyes for approximately 1 week.
  Arms: CSF-1 Component #1
Drug: CSF-1 Component #2 — This treatment arm consists of a single concentration of CSF-1 Component #2. Subjects randomized to the CSF-1 Component #2 treatment arm will receive their first dose of CSF-1 Component #2 in-office at Visit 2. All subjects will dose twice a day in both eyes with a single drop for approximately 1 week. At Visit 3, subjects randomized to the CSF-1 Component #2 arm will continue dosing with the same concentration of CSF-1 Component #2. Subjects will continue dosing twice a day in both eyes for approximately 1 week.
  Arms: CSF-1 Component #2

SUMMARY:
This is a 4-visit, multi-center, randomized, double-masked, parallel group study evaluating the safety and efficacy of CSF-1 in the treatment of presbyopia.

DETAILED DESCRIPTION:
This is a 4-visit, multi-center, randomized, double-masked, parallel group study evaluating the safety and efficacy of CSF-1 in the treatment of presbyopia. Approximately 150 subjects will be enrolled across 7 study centers in the United States. At Visit 2, subjects will be randomized 1:1:1 to one of three treatment arms: CSF-1, CSF-1 Component #1, or CSF-1 Component #2. All subjects will dose twice a day in both eyes with a single drop of their assigned treatment for approximately 1 week. At Visit 3, subjects randomized to CSF-1 will now receive a different concentration of CSF-1, subjects randomized to CSF-1 Component #1 will receive a different concentration of CSF-1 Component #1 and subjects randomized to CSF-1 Component #2 will continue dosing with the same concentration of CSF-1 Component #2. All subjects will continue dosing twice a day in both eyes for approximately 1 week.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must:

  1. Have presbyopia

Exclusion Criteria:

* Subjects must not:

  1. Have any contraindications to the study medications or diagnoses that would confound the study data

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 166 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Orasis Investigative Site, Newport Beach, California
  - Orasis Investigative Site, Littleton, Colorado
  - Orasis Investigative Site, Andover, Massachusetts
  - Orasis Investigative Site, Bloomington, Minnesota
  - Orasis Investigative Site, Cranberry Township, Pennsylvania
  - Orasis Investigative Site, Memphis, Tennessee
  - Orasis Investigative Site, Draper, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CSF-1-FDC: pilocarpine HCl + diclofenac Na (fixed dose combination), 1 drop in each eye administered 2 times a day
- Pilo: pilocarpine HCl (alone), 1 drop in each eye administered 2 times a day
- Diclo: diclofenac Na (serves as control group), 1 drop in each eye administered 2 times a day
Period: Overall Study
Arm/Group | CSF-1-FDC | Pilo | Diclo
Started | 53 | 55 | 58
Completed | 52 | 52 | 57
Not Completed | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- CSF-1-FDC: pilocarpine HCl + diclofenac Na (fixed dose combination)
- Pilo: pilocarpine HCl (alone)
- Diclo: diclofenac Na (serves as control group)
- Total: Total of all reporting groups
Arm/Group | CSF-1-FDC | Pilo | Diclo | Total
Number analyzed (Participants) | 53 | 55 | 58 | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (3.96) | 54.9 (4.93) | 54.1 (4.94) | 54.6 (4.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 39 | 33 | 102
  Male | 23 | 16 | 25 | 64
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2 | 4
  Not Hispanic or Latino | 52 | 54 | 56 | 162
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 9 | 7 | 26
  White | 41 | 45 | 48 | 134
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 53 | 55 | 58 | 166

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With ≥ 3 Lines Gain in Near Best Distance Corrected Visual Acuity (BDCVA) (at 40 cm)
Description: Number of subjects with a ≥ 3-line gain in near BDCVA (at 40 cm) at 1 hour post dose after 1 week treatment with CSF-1-Fixed Dose Combination (FDC) low dose (pilocarpine HCl 0.2% + diclofenac 0.006%) or pilocarpine HCl 0.2% alone or diclofenac 0.006% alone
Time Frame: 1 hour post dose on day 8
Population: The primary analysis was conducted on the per protocol (PP) study population set and therefore the number of subjects is slightly different than from the overall participant flow.
Measure: Count of Participants; unit: Participants
Arm/Group | CSF-1-FDC | Pilo | Diclo
Number analyzed (Participants) | 51 | 50 | 56
Participants | 10 | 12 | 10
Statistical Analysis 1: Comparison: CSF-1-FDC vs Diclo; This analysis relates to Day 8 up to when pilocarpine HCl 0.2% either in CSF-1-FDC or as pilocarpine alone was administered for one week; Test type: Superiority; p = 0.8445, Regression, Logistic; Odds Ratio (OR) = 1.103, 95% CI 2-sided [0.413 to 2.949]
Statistical Analysis 2: Comparison: Pilo vs Diclo; Test type: Superiority; p = 0.2660, Regression, Logistic; Odds Ratio (OR) = 1.646, 95% CI 2-sided [0.684 to 3.958]

2. Primary Outcome: Number of Subjects With ≥ 3 Lines Gain in BDCVA (at 40 cm)
Description: Number of subjects with a ≥ 3-line gain in near BDCVA (at 40 cm) at 1 hour post dose after 1 week treatment with CSF-1-FDC (pilocarpine HCl 0.4% + diclofenac 0.006%) or pilocarpine HCl 0.4% alone or diclofenac 0.006% alone
Time Frame: 1 hour post dose on day 15
Population: The primary analysis was conducted on the per protocol (PP) study population set and therefore the number of subjects is slightly different than from the overall participants flow.
Measure: Count of Participants; unit: Participants
Arm/Group | CSF-1-FDC | Pilo | Diclo
Number analyzed (Participants) | 51 | 49 | 56
Participants | 22 | 23 | 9
Statistical Analysis 1: Comparison: CSF-1-FDC vs Diclo; Test type: Superiority; p = 0.0015, Regression, Logistic; Odds Ratio (OR) = 3.664, 95% CI 2-sided [1.646 to 8.154]
Statistical Analysis 2: Comparison: Pilo vs Diclo; Test type: Superiority; p = 0.0002, Regression, Logistic; Odds Ratio (OR) = 4.745, 95% CI 2-sided [2.088 to 10.786]

3. Secondary Outcome: Number of Subjects With ≥ 2 Lines Gain in BDCVA (at 40 cm)
Description: Number of subjects with a ≥ 2-line gain in near BDCVA (at 40 cm0 at 1 hour post dose after 1 week treatment with CSF-1-FDC (pilocarpine HCl 0.2% + diclofenac 0.006%) or pilocarpine HCl 0.2% alone or diclofenac 0.006% alone
Time Frame: 1 hour post dose on day 8
Population: The analysis was conducted on the per protocol (PP) study population set and therefore the number of subjects is slightly different than from the overall participants flow.
Measure: Count of Participants; unit: Participants
Arm/Group | CSF-1-FDC | Pilo | Diclo
Number analyzed (Participants) | 51 | 50 | 56
Participants | 24 | 25 | 18
Statistical Analysis 1: Comparison: CSF-1-FDC vs Diclo; Test type: Superiority; p = 0.1145, Chi-squared
Statistical Analysis 2: Comparison: Pilo vs Diclo; Test type: Superiority; p = 0.0616, Chi-squared

4. Secondary Outcome: Number of Subjects With ≥ 2 Lines Gain in BDCVA (at 40 cm)
Description: Number of subjects with a ≥ 2-line gain in near BDCVA (at 40 cm) at 1 hour post dose after 1 week treatment with CSF-1-FDC (pilocarpine HCl 0.4% + diclofenac 0.006%) or pilocarpine HCl 0.4% alone or diclofenac 0.006% alone
Time Frame: 1 hour post dose on day 15
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | CSF-1-FDC | Pilo | Diclo
Number analyzed (Participants) | 51 | 49 | 56
Participants | 35 | 39 | 24
Statistical Analysis 1: Comparison: CSF-1-FDC vs Diclo; Test type: Superiority; p = 0.0074, Chi-squared
Statistical Analysis 2: Comparison: Pilo vs Diclo; Test type: Superiority; p = 0.0001, Chi-squared

ADVERSE EVENTS:
Time Frame: During the 2 weeks duration of the study.
Description: Treatment emergent adverse events (TEAEs) reported, elicited, and observed during clinical visits. In the CSF-1-FDC and the pilocarpine alone groups, TEAEs are reported for both doses of pilocarpine, as no separate analysis for TEAEs reported on Day 8 and Day 15 was planned in the protocol or statistical analysis plan.
Arm/Group | CSF-1-FDC | Pilo | Diclo
All-Cause Mortality (participants affected / at risk) | 0/53 | 1/55 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/53 | 1/55 | 0/58
Other Adverse Events (participants affected / at risk) | 10/53 | 13/55 | 6/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CSF-1-FDC (N=53) | Pilo (N=55) | Diclo (N=58)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — The subject experienced a non-ocular SAE of coronary artery disease which resulted in death. The SAE was severe and considered by the investigator to be not related to the study drug.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CSF-1-FDC (N=53) | Pilo (N=55) | Diclo (N=58)
Conjunctival hyperemia (Eye disorders) | 3 | 2 | 0
Vision blurred (Eye disorders) | 1 | 6 | 3
Instillation site pain (General disorders) | 5 | 3 | 2
Headache (Nervous system disorders) | 1 | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-06-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT03885011/Prot_000.pdf
  • Statistical Analysis Plan (2019-07-24): https://cdn.clinicaltrials.gov/large-docs/11/NCT03885011/SAP_001.pdf